CLINICAL TRIAL: NCT07164664
Title: External Oblique Intercostal Block Versus Port-Site Infiltration for Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: External Oblique Intercostal Block in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra Turunc, Director, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EOIBLIALC2025
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Pain, Acute; Opioid Use
Keywords: Postoperative pain; regional anesthesia; external oblique intercostal block
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer (Urbaniak and Plous, 2013)'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based "Research Randomizer" (Urbaniak and Plous 2013) tool to give each participation number to a random group with a 1:1 ratio. A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist administering the block/blocks about which group the patient is in immediately before administration. Researchers, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EOIB (Active Comparator): A bilateral External Oblique Intercostal Block (30 ml, %0.25 bupivacaine, bilaterally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: External Oblique Intercostal Block; Drug: ıv morphine PCA
- Group PSI (Active Comparator): Port sites injection (5 mL at each port site, 0.25% bupivacaine solution ) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Port-Site Infiltration; Drug: ıv morphine PCA

INTERVENTIONS:
Procedure: External Oblique Intercostal Block — Bilateral ultrasound-guided External Oblique Intercostal Block (30 mL, 0.25% bupivacaine, bilaterally) will be performed. All patients will receive multimodal analgesia, including a single dose of IV tenoxicam 20 mg. Additionally, 15 mg/kg IV paracetamol (based on IBW) will be administered at skin closure and continued every 6 hours postoperatively. A standardized IV PCA protocol will be initiated using a PCA device programmed to deliver morphine boluses of 0.01-0.015 mg/kg (IBW), with a 6-minute lockout and a 4-hour maximum of 0.1-0.15 mg/kg (IBW). Upon arrival in the PACU, patients with a resting NRS ≥4 will receive titrated IV morphine boluses of 0.03 mg/kg (IBW; max 10 mg) every 10 minutes until pain is controlled. In the surgical ward, patients with breakthrough pain (NRS ≥4) despite PCA use will receive IV tramadol 1-1.5 mg/kg (IBW) in 50-100 mg slow doses, not exceeding 400 mg/day.All patients will receive 8 mg dexamethasone and 0.15 mg/kg ondansetron (IBW) for PONV prophylaxis.
  Other Names: EOIB
  Arms: Group EOIB
Procedure: Port-Site Infiltration — Before port placement, 0.25% bupivacaine solution will be injected into the laparoscopic port insertion sites (5 mL at each port site).
  Other Names: PSI
  Arms: Group PSI
Drug: ıv morphine PCA — A standardized IV PCA protocol will be initiated for all patients using a PCA device (Body Guard 575 pain manager, UK), programmed to deliver morphine boluses of 0.01-0.015 mg/kg (IBW), with a 6-minute lockout and a 4-hour maximum dose of 0.1-0.15 mg/ kg (IBW). No basal infusion will be used.
  Other Names: PCA

SUMMARY:
Adequate postoperative pain management is essential for improving patient comfort and recovery after laparoscopic cholecystectomy. This study evaluated the effectiveness of the external oblique intercostal block compared with port-site infiltration in terms of pain scores and opioid consumption during the first 24 hours after surgery.

DETAILED DESCRIPTION:
Adequate pain relief in the postoperative period is a crucial determinant of patient comfort, early mobilization, and overall recovery after laparoscopic cholecystectomy. Effective analgesia not only improves patient satisfaction but also reduces postoperative complications, facilitates respiratory function, and shortens hospital stay. Conversely, insufficient pain control may lead to undesirable outcomes such as delayed mobilization, nausea, vomiting, increased opioid requirements, and prolonged recovery.

Regional anesthesia techniques, particularly abdominal wall and fascial plane blocks, have gained increasing attention as part of multimodal analgesia strategies aimed at reducing opioid consumption and minimizing related adverse effects. Among these, the external oblique intercostal block (EOIB) has recently been described as a novel regional technique that may provide effective postoperative pain relief.

In clinical practice, port-site infiltration with local anesthetics is a commonly used and simple technique for providing postoperative analgesia in laparoscopic procedures, although its effectiveness may be limited.

The present study was designed to compare the effectiveness of the external oblique intercostal block with port-site infiltration in patients undergoing laparoscopic cholecystectomy, with a focus on postoperative pain scores and opioid consumption during the first 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 undergoing elective Laparoscopic Cholecystectomy
* American Society of Anesthesiologists (ASA)classification I-III patients.
* Patients who can use PCA.
* Patients who will sign the informed consent form.

Exclusion Criteria:

* They will refuse to participate.
* They will have a body mass index (BMI) greater than 35 kg/m2.
* They will have contraindications to peripheral nerve blocks (e.g., coagulopathy, abnormal INR, thrombocytopenia, local or systemic infection).
* They will have clinically significant cardiovascular or cerebrovascular disease.
* They will have severe hepatic, renal, or respiratory dysfunction. They will have known drug allergies.
* They will have a history of substance abuse.
* They will have chronic opioid use, defined as regular use of ≥15 mg oral morphine equivalent per day for at least 30 consecutive days within the past 3 months.
* They will have chronic pain syndromes (e.g., fibromyalgia, diabetic neuropathy, or chronic low back pain).
* They will have neuropsychiatric disorders or cognitive impairment that precludes effective communication with the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | Postoperative day 1
  The primary outcome will be defined as cumulative opioid consumption during the first 24 hours following surgery, which will be calculated in intravenous morphine milligram equivalents (IV-MME), encompassing both PCA- administered morphine and rescue intravenous tramadol, according to the standardized ESAIC conversion guidelines. Patients can request opioids via a PCA device when their NRS score is≥ 4.

SECONDARY OUTCOMES:
Cumulative opioid consumption in the first 12 hours after surgery | Postoperative 12 hours
  The secondary outcome will be defined as cumulative opioid consumption during the first 12 hours following surgery, calculated in intravenous morphine milligram equivalents (IV-MME). This will include both PCA-administered morphine and rescue intravenous tramadol, in accordance with the standardized ESAIC conversion guidelines. Patients may request opioids using a PCA device when their NRS score is ≥ 4.
Intraoperative Remifentanil Consumption | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 150 minutes
  Total intraoperative remifentanil consumption will be recorded in micrograms (μg) from the start of anesthesia induction until the end of surgery.
Numerical Rating Scale Assessment of Postoperative Pain | Postoperative day 1
  Pain scores will be assessed using the 11-point Numerical Rating Scale (NRS), where 0 indicates no pain and 10 represents the worst imaginable pain. Evaluations will be performed both at rest (static) and during coughing or deep breathing (dynamic). Assessments will be conducted in the post-anesthesia care unit (PACU) after extubation and once communication is established, and subsequently at 3, 6, 12 and 24 hours postoperatively.
Time to First Opioid Demand via PCA | Postoperative day 1
  Defined as the time elapsed from the patient's arrival in the post-anesthesia care unit (PACU) to the first patient- initiated opioid request via the patient-controlled analgesia (PCA) device.
The number of patients who required rescue analgesia. | Postoperative day 1
  The number of patients who required additional IV tramadol due to breakthrough pain (NRS ≥4) despite PCA use.
The patient number of Rescue antiemetic Requirement | Postoperative day 1
  All patients received standard prophylaxis for postoperative nausea and vomiting (PONV), including 8 mg IV dexamethasone before induction and 0.15 mg/kg IV ondansetron (based on ideal body weight) approximately 20 minutes before the end of surgery. PONV was assessed at 0, 3, 6, 12, 18, and 24 hours after extubation using a 5- point scale (0 = no nausea to 4 = multiple episodes of vomiting). Patients with a PONV score ≥3 received rescue treatment with 10 mg IV metoclopramide in 100 mL normal saline via slow infusion. The number of patients requiring rescue antiemetic therapy was recorded.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients has any complications -directly related to the block or the drug used in the block- will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Esra Turunc, Study Director — Ondokuz Mayis University, School of Medicine, Department of Anesthesiology
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)